CLINICAL TRIAL: NCT01487759
Title: Metabolite Profiling of the Impact of Oligofructose Enriched Inulin in Crohn's Disease Patients
Brief Title: Prebiotic Effect on Metabolites in Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Principal investigator, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: ML4789
Record Dates: First submitted 2011-12-06; First posted 2011-12-07 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prebiotic (Active Comparator)
  Interventions: Dietary Supplement: Oligofructose enriched inulin
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Oligofructose enriched inulin
  Arms: Prebiotic
Dietary Supplement: Maltodextrin
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the influence of the prebiotic oligofructose enriched inulin on the metabolite pattern in Crohn's disease patients.

ELIGIBILITY:
Inclusion Criteria:

* crohn's disease

Exclusion Criteria:

* severe crohn's disease (harvey bradshaw index >12)
* pregnancy
* history of colectomy
* use of antibiotics 4-wks before start of the study
* use of sulfapyridine
* use of commercially available prebiotics and probiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-03; Study Completion 2009-07

CONTACTS AND LOCATIONS:
Locations (1):
- KULeuven, Leuven, Belgium